CLINICAL TRIAL: NCT05006872
Title: Supporting People With Type 2 Diabetes in Effective Use of Their Medicine Through a System Comprising Mobile Health Technology Integrated With Clinical Care
Brief Title: mHealth Intervention to Support Diabetes Medication Adherence
Acronym: DIABE-TEXT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RTI2018-096935-A-100_rct; IB 4320/20 PI (Other: Research Ethics Committee of the Balearic Islands)
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; medication; adherence; glycaemic control; healthy lifestyle; mHealth; SMS
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Healthcare providers (doctors and nurses from the participants' health centres, do not know if their patients are participating in the study nor the group (intervention vs control) they are. Just if a patient ask them for more information related to the study or text messages, they will know about it. Also, the interviewers that evaluate and register participants data are masked until randomization. After 12 months of follow-up, the interviewers will be masked before post-intervention evaluation. The primary outcome HbA1c is an objective measure and assessors of this outcome will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DIABE-TEXT (Experimental): Participants allocated to the intervention group will receive text messages in their mobile phones with content about diabetes management, general information about diabetes, medicines, diet and physical activity recommendations and motivational prompts to engage participants in a healthy lifestyle and a good adherence to medication plan. They will also receive reminders for healthcare visits, drug dispensation from the pharmacy and updated results from blood test records.
  Interventions: Device: DIABE-TEXT
- Usual care (No Intervention): Participants allocated to the control group will not receive any intervention apart from usual care.

INTERVENTIONS:
Device: DIABE-TEXT — Participants will receive 170 text messages in their mobile phones during twelve months.
  Arms: DIABE-TEXT

SUMMARY:
This study aims at evaluating the effectiveness of an intervention based on the use of a mobile-device based system delivering automated, tailored brief text messages to offer support for medicine use and lifestyle recommendations alongside usual care to people with type 2 diabetes.

DETAILED DESCRIPTION:
A list of patients registered in primary care centers of the Balearic Islands and potentially meeting the eligibility criteria will be obtained from electronic health records (EHRs). A research assistant will contact the potential participants via phone to invite them to the study and confirm eligibility. All eligible participants will complete informed consent followed by baseline assessment over the phone before randomization. Participants will be randomly allocated using a computer-generated randomization sequence. All participants will continue with their usual diabetes care including all medical visits, tests, and diabetes support programs throughout the study. In addition, the intervention group will receive the text messaging intervention. Control participants will receive usual care only.

After twelve months of follow-up, all participants will complete post-intervention assessments via phone interview. Data on glycemic control (HbA1c) at baseline and post-intervention will be extracted from EHRs, as according to the protocol used for primary care providers in the Balearic Islands, patients with poor glycemic control (HbA1c >8% ) must request an HbA1c determination every six months. Results of the most recent determination will be extracted from electronic medical records. For those patients with no recorded HbA1c within the previous four months, the research assistant will contact the primary care center to arrange blood test analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients registered in the Public Health Service of the Balearic Islands
* With type 2 diabetes
* At least one prescription of a glucose-lowering drug
* With results of HbA1c>8% from 6 months prior to recruitment

Exclusion Criteria:

* Younger than 18 years old
* With insulin treatment
* Participating in another research study
* Not living in the Balearic Islands at some point during the study development

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 742 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ignacio Ricci-Cabello, Palma de Mallorca, Balearic Islands, Spain

REFERENCES:
- [Background] Zamanillo-Campos R, Fiol-DeRoque MA, Serrano-Ripoll MJ, Mira-Martinez S, Llobera-Canaves J, Taltavull-Aparicio JM, Leiva-Rus A, Ripoll-Amengual J, Angullo-Martinez E, Socias-Buades IM, Masmiquel-Comas L, Konieczna J, Zaforteza-Dezcallar M, Boronat-Moreiro MA, Gervilla-Garcia E, Ricci-Cabello I. DiabeText, a mobile health intervention to support medication taking and healthy lifestyle in adults with type 2 diabetes: Study protocol for a randomized controlled trial. Contemp Clin Trials. 2024 Jan;136:107399. doi: 10.1016/j.cct.2023.107399. Epub 2023 Nov 22. PMID 37995967

RESULTS

PARTICIPANT FLOW:
Groups:
- DIABE-TEXT: Participants allocated to the intervention group received 167 text messages in their mobile phones with content about diabetes management, general information about diabetes, medicines, diet and physical activity recommendations and motivational prompts to engage participants in a healthy lifestyle and a good adherence to medication plan. They also received reminders for healthcare visits, drug dispensation from the pharmacy and updated results from blood test records.
  DIABE-TEXT: Participants will receive 170 text messages in their mobile phones during twelve months.
- Usual Care: Participants allocated to the control group did not receive any intervention apart from usual care.
Period: Overall Study
Arm/Group | DIABE-TEXT | Usual Care
Started | 371 | 371
Completed | 334 | 340
Not Completed | 37 | 31
Not completed — Lost to Follow-up | 37 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DIABE-TEXT | Usual Care | Total
Number analyzed (Participants) | 371 | 371 | 742
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10) | 65 (10) | 65 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 154 | 309
  Male | 216 | 217 | 433
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 371 | 371 | 742
Glycated hemoglobin (HbA1c) [Median (Inter-Quartile Range); unit: Percentage of HbA1c] | 8.1 [7.7 to 8.7] | 8.0 [7.6 to 8.8] | 8.1 [7.7 to 8.8]

OUTCOME MEASURES:

1. Primary Outcome: Glycated Hemoglobin (HbA1c) (%)
Description: HbA1c was extracted as percentage which is calculated following the standard formulae [HbA1c(%)=(HbA1c(mmol/mol)+23.5)/ 10.93] based on its concentration in blood samples. It identifies average plasma glucose concentration (1).
  The most recent HbA1c data registered between 6th of April and 12th of November in 2021 were extracted for all participants at baseline.
  At post-intervention, we extracted the most recent data which was available between 21st September 2022 and 21st February 2023.
Time Frame: Baseline and post-intervention at 12 months
Population: The number analyzed post-intervention differs from overall number analyzed because of losses to follow-up.
Measure: Median (Inter-Quartile Range); unit: Percentage of HbA1c
Arm/Group | DIABE-TEXT | Usual Care
Number analyzed (Participants) | 371 | 371
Percentage of HbA1c
  Baseline | 8.1 [7.7 to 8.7] | 8.0 [7.6 to 8.8]
  Post-intervention: number analyzed (Participants) | 309 | 321
  Post-intervention | 7.5 [6.7 to 8.2] | 7.4 [6.7 to 8.3]

2. Primary Outcome: Mean Adherence to Antidiabetic Drugs (%)
Description: We calculated adherence in terms of medication possession ratio (MPR), defined as the number of days with treatment as medication being dispensed from the pharmacy to the patient (numerator), out of the total days of treatment prescribed by the doctor (denominator) (2):
  MPR = [Days with treatment (prescription dispensed) / Days with treatment as prescribed by the doctor] x 100
  At baseline it was calculated as the mean adherence for all the glucose lowering drugs prescribed during the 6 months previous to recruitment excluding insulin.
  At post-intervention it was calculated as the mean adherence for all the glucose lowering drugs prescribed during the 12 months follow-up excluding insulin.
Time Frame: Baseline and post-intervention at 12 months
Measure: Median (Inter-Quartile Range); unit: Medication possession ratio (percentage)
Arm/Group | DIABE-TEXT | Usual Care
Number analyzed (Participants) | 371 | 371
Medication possession ratio (percentage)
  Baseline | 95.1 [81.8 to 99.3] | 96.2 [83.1 to 99.3]
  Post-intervention | 90.4 [76.2 to 97.7] | 91.0 [73.6 to 97.8]

3. Secondary Outcome: Number of Participants Classified as Adherent Based on Self-reported Adherence to Antidiabetic Medication (7 Items ad Hoc Questionnaire)
Description: Number of participants classified as adherent based on Self-reported adherence to glucose medications was measured with a 7-items ad hoc questionnaire adapted from Chaves-Torres et al. for people with type 2 diabetes. Participants who obtained 7 points were considered adherent while the ones with < 7 points were non-adherent.
Time Frame: Baseline and post-intervention at 12 months
Population: The number analyzed post-intervention differs from overall number analyzed at baseline because of lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | DIABE-TEXT | Usual Care
Number analyzed (Participants) | 371 | 371
Participants
  Baseline | 205 | 194
  Post-intervention: number analyzed (Participants) | 334 | 340
  Post-intervention | 220 | 197

4. Secondary Outcome: Health-related Quality of Life (EQ-5D-5L)
Description: The 5-level EuroQol 5-dimensional questionnaire (EQ-5D-5L) questionnaire was completed at baseline and post-intervention interviews. The index score was calculated using STATA syntax code and values with the Spanish value set according to Ramos-Goñi JM et al. Information about the EQ-5D index, derived using a value set, can be presented in much the same way as the EQ VAS data, i.e. using measures of central tendency and dispersion, such as mean values and the SD (or standard error). If the data are skewed, the median values and the 25th and 75th percentiles could be presented. Note, when reporting index values, a maximum of three decimal places is usually sufficient. Index values can range between 0 to 1. Higher EQ-5D index scores mean better quality of life related to health status.
Time Frame: Baseline and post-intervention at 12 months
Population: The number analyzed post-intervention differs from overall number analyzed at baseline because of lost to follow-up.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | DIABE-TEXT | Usual Care
Number analyzed (Participants) | 371 | 371
score on a scale
  Baseline | 0.93 [0.88 to 1] | 0.93 [0.89 to 1]
  Post-intervention: number analyzed (Participants) | 334 | 340
  Post-intervention | 1 [0.92 to 1] | 0.97 [0.89 to 1]

5. Secondary Outcome: Self-efficacy to Manage Diabetes (DSES-S)
Description: The validated scale known as diabetes management self-efficacy scale in Spanish (DSES-S) was completed at baseline and post-intervention interviews. The scales consist of 8 Likert-type 10-point items. The score for each item was the number circled. If two consecutive numbers were circled, the lower number (less self-efficacy) was coded. If the numbers were not consecutive, the item was not scored. The final score for the scale is the mean of the eight items (points). Therefore, DSES-S scores range between 1 to 10. If more than two items were missing, we did not score the scale following instructions. Higher number indicates higher self-efficacy.
Time Frame: Baseline and post-intervention at 12 months
Population: The number analyzed post-intervention differs from overall number analyzed at baseline because of lost to follow-up.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | DIABE-TEXT | Usual Care
Number analyzed (Participants) | 371 | 371
score on a scale
  Baseline | 6.9 [5.8 to 8.0] | 6.9 [5.9 to 7.9]
  Post-intervention: number analyzed (Participants) | 334 | 340
  Post-intervention | 8.6 [7.4 to 9.3] | 8.0 [6.6 to 8.9]

6. Other Pre Specified Outcome: 14-point Mediterranean Diet Adherence Screener (MEDAS-14)
Description: The 14-point Mediterranean Diet Adherence Screener (MEDAS-14) questionnaire was registered at baseline and post-intervention. Participants were classified as low adherents (≤5), moderate adherents (6 to 9 points) or high adherents (≥10 points) according to the results obtained that can range between 1 to 14 points. After that, we joined moderate adherents with high adherents and tagged them as adherents to the Mediterranean Diet, while low adherents were considered non-adherents to the Mediterranean diet. Therefore, we presented the number of participants adherent to the Mediterranean Diet.
Time Frame: Baseline and post-intervention at 12 months
Population: The number analyzed post-intervention differs from overall number analyzed at baseline because of lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | DIABE-TEXT | Usual Care
Number analyzed (Participants) | 371 | 371
Participants
  Baseline | 271 | 281
  Post-intervention: number analyzed (Participants) | 334 | 340
  Post-intervention | 171 | 169

7. Other Pre Specified Outcome: International Physical Activity Questionnaire (IPAQ)
Description: A 6-items adapted from the short version of the International Physical Activity Questionnaire (IPAQ) (11) was registered at baseline and post-intervention. Participants were classified as having a low, moderate or high level of physical activity based on metabolic equivalent of task (METs) calculation. After that, we joined the participants that presented moderate or high level of physical activity and tagged them as adherents to Physical Activity recommendations, while low levels of Physical Activity was considered as being non-adherent to the Physical Activity Recommendations. Therefore, we presented the number of participants adherent to the Physical Activity Recommendations.
Time Frame: Baseline and post-intervention at 12 months
Population: The number analyzed post-intervention differs from overall number analyzed at baseline because of lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | DIABE-TEXT | Usual Care
Number analyzed (Participants) | 371 | 371
Participants
  Baseline | 240 | 245
  Post-intervention: number analyzed (Participants) | 334 | 340
  Post-intervention | 171 | 194

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at 12-months post-intervention
Description: Serious adverse events were not assessed; therefore, the number of affected participants cannot be reported accurately.
Arm/Group | DIABE-TEXT | Usual Care
All-Cause Mortality (participants affected / at risk) | 6/371 | 2/371
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 2/371 | 0/371
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DIABE-TEXT (N=371) | Usual Care (N=371)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
1. Difficulties in accurately measuring participant adherence due to message comprehension uncertainties and relay through caregivers, potentially diluting intervention reach.
2. Lack of intermediate evaluations during follow-up.
3. Lack of registration of social variables.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/72/NCT05006872/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/72/NCT05006872/ICF_001.pdf